CLINICAL TRIAL: NCT05724693
Title: A Phase 1, Multicenter, Open-Label, Parallel-Group, Pharmacokinetic Single Dose Study of Bemnifosbuvir (AT-527) in Adult Subjects With Normal and Impaired Hepatic Function
Brief Title: Study of Bemnifosbuvir in Subjects With Normal and Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT-03A-010
Record Dates: First submitted 2023-01-24; First posted 2023-02-13 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteer; Hepatic Impairment
MeSH Terms: interventions — AT-511

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 1 -Mild Hepatic Impairment (Experimental): Drug: single dose Bemnifosbuvir (BEM)
  Interventions: Drug: Bemnifosbuvir (BEM)
- Group 2-Moderate Hepatic Impairment (Experimental): Drug: single dose Bemnifosbuvir (BEM)
  Interventions: Drug: Bemnifosbuvir (BEM)
- Group 3 - Healthy Subjects matching mild and moderate impairment groups (Experimental): Drug: single dose Bemnifosbuvir (BEM)
  Interventions: Drug: Bemnifosbuvir (BEM)
- Group 4 - Severe Hepatic Impairment (Experimental): Drug: single dose Bemnifosbuvir (BEM)
  Interventions: Drug: Bemnifosbuvir (BEM)
- Group 5 - Normal hepatic function matching severe impairment group (Experimental): Drug: single dose Bemnifosbuvir (BEM)
  Interventions: Drug: Bemnifosbuvir (BEM)

INTERVENTIONS:
Drug: Bemnifosbuvir (BEM) — Day 1: A single dose of BEM will be administered
  Other Names: AT-527

SUMMARY:
To Assess the Effect of Hepatic Impairment on the Pharmacokinetics of Bemnifosbuvir After a Single Dose

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug
* Females must have a negative pregnancy test at Screening and prior to dosing
* BMI of 18.5 to 42.0 kg/m2
* Willing to comply with the study requirements and to provide written informed consent

Subjects with Normal Hepatic Function (Groups 3 and 5):

* Medically healthy, in the opinion of an Investigator
* Must match by gender, age (± 10 years), and BMI (± 20%) to the pooled mean values of subjects with hepatic impairment

Hepatic Impaired Subjects (Groups 1, 2, and 4):

* Considered stable for at least 1 month prior to Screening, as per the judgement of an Investigator
* When applicable, presence of mild hepatic impairment (Child-Pugh Class A: score of 5 to 6), moderate hepatic impairment (Child-Pugh Class B: score of 7 to 9) or severe hepatic impairment (Child-Pugh Class C: score of 10 to 15). Hepatic impairment should be stable for at least 1 month prior to Screening

Exclusion Criteria:

* Pregnant or breastfeeding
* Infected with hepatitis B virus, hepatitis C virus, HIV or COVID-19
* Abuse of alcohol or drugs
* Use of other investigational drugs within 28 days of dosing
* Other clinically significant medical conditions or laboratory abnormalities

Hepatic Impaired Subjects (Groups 1, 2, and 4):

* Currently undergoing any method of dialysis
* History of liver transplant
* Presence of poorly controlled Type 1 or Type 2 diabetes as defined by Hemoglobin A1c (HbA1c) > 10%
* Evidence of hepatic carcinoma presence at Screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of BEM Maximum plasma concentration (Cmax) | Day 1
Pharmacokinetics (PK) of BEM Area under the plasma concentration-time curve (AUC) | Day 1
Pharmacokinetics (PK) of BEM AUC | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site Orlando Clinical Research Center, Orlando, Florida, United States